CLINICAL TRIAL: NCT01085760
Title: A Pilot Study of Vancomycin or Metronidazole in Patients With Primary Sclerosing Cholangitis
Acronym: PSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: PSC Partners Seeking a Cure (Other)
Responsible Party: Principal Investigator, Jayant A. Talwalkar, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-008247
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Results first posted 2013-09-19 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-07

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Vancomycin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vancomycin 125 mg orally 4 times a day (Experimental): The patients will be randomized into four groups of ten patients: one group will receive low dose vancomycin, one group will receive high dose vancomycin, one group will receive low dose metronidazole and one group will receive high dose metronidazole.
  Interventions: Drug: Vancomycin
- Vancomycin 250 mg orally 4 times a day (Experimental)
  Interventions: Drug: Vancomycin
- Metronidazole 250 mg orally 3 times a day (Experimental)
  Interventions: Drug: Metronidazole
- Metronidazole 500 mg orally 3 times a day (Experimental)
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Vancomycin — Comparison of different doses of drug
  Arms: Vancomycin 125 mg orally 4 times a day
Drug: Vancomycin — Comparison of different doses of drug
  Arms: Vancomycin 250 mg orally 4 times a day
Drug: Metronidazole — Comparison of different doses of drug
  Arms: Metronidazole 250 mg orally 3 times a day
Drug: Metronidazole — Comparison of different doses of drug
  Arms: Metronidazole 500 mg orally 3 times a day
Drug: Vancomycin — Comparison of different drug doses
  Arms: Vancomycin 125 mg orally 4 times a day

SUMMARY:
The purpose of this study is to determine whether Vancomycin or Metronidazole is safe and beneficial in the treatment of Primary Sclerosing Cholangitis.

DETAILED DESCRIPTION:
In this protocol, we propose the assessment of potential beneficial effects of the antibiotics vancomycin and metronidazole on liver biochemistries, liver related symptoms and Mayo risk score in patients with PSC. The patients will be randomized into four groups of ten patients: one group will receive low dose vancomycin, one group will receive high dose vancomycin, one group will receive low dose metronidazole and one group will receive high dose metronidazole. Each group will be treated for three months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PSC established by alkaline phosphatase >1.5 times and/or two fold elevation of liver transaminases (AST and/or ALT) for at least 6 months duration.
* Cholangiography demonstrating intrahepatic and/or extrahepatic biliary obstruction, beading, or narrowing consistent with PSC.
* Both genders.
* Age ≥ 18 years old and < than 75 years old.
* Patient's informed consent for study participation.

Exclusion Criteria:

* Treatment with systematic antibiotics, azulfidine, ursodeoxycholic acid, corticosteroids, colchicine, methotrexate, azathioprine, cyclosporine, chlorambucil, budesonide, pentoxifylline, tacrolimus, silymarin or prednisone in the preceding three months.
* Active drug or alcohol use.
* Prior history of allergic reactions to the antibiotics which will be used in the study.
* Any condition that, in the opinion of the investigator, would interfere with the patients' ability to complete the study safely or successfully.
* Evidence of decompensated liver disease such as recurrent variceal bleeding, refractory ascites or spontaneous hepatic encephalopathy.
* Anticipated need for transplantation in one year (Mayo survival model <80% one-year survival without transplant).
* Findings highly suggestive of liver disease of other etiology such as chronic alcoholic liver disease, chronic hepatitis B or C infection, hemochromatosis, Wilson's disease, 1-antitrypsin deficiency, non-alcoholic steatohepatitis, primary biliary cirrhosis or secondary sclerosing cholangitis.
* Pregnancy or current lactation. Subjects becoming pregnant during the study will be withdrawn.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayant A Talwalkar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Tabibian JH, Weeding E, Jorgensen RA, Petz JL, Keach JC, Talwalkar JA, Lindor KD. Randomised clinical trial: vancomycin or metronidazole in patients with primary sclerosing cholangitis - a pilot study. Aliment Pharmacol Ther. 2013 Mar;37(6):604-12. doi: 10.1111/apt.12232. Epub 2013 Feb 5. PMID 23384404

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 adult patients with primary sclerosing cholangitis (PSC) were enrolled between February 2010 and November 2011 at Mayo Clinic, Rochester MN.
Groups:
- Low Dose Vancomycin: Vancomycin 125 mg 4 times a day
- High Dose Vancomycin: Vancomycin 250 mg 4 times a day
- Low Dose Metronidazole: Metronidazole 250 mg 3 times a day
- High Dose Metronidazole: metronidazole 500 mg 3 times a day
Period: Overall Study
Arm/Group | Low Dose Vancomycin | High Dose Vancomycin | Low Dose Metronidazole | High Dose Metronidazole
Started | 8 | 9 | 9 | 9
Completed | 7 | 8 | 7 | 6
Not Completed | 1 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Vancomycin | High Dose Vancomycin | Low Dose Metronidazole | High Dose Metronidazole | Total
Number analyzed (Participants) | 8 | 9 | 9 | 9 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 9 | 9 | 32
  >=65 years | 0 | 3 | 0 | 0 | 3
Age Continuous [Median (Full Range); unit: years] | 40 [20 to 60] | 42 [27 to 70] | 35 [21 to 64] | 40 [20 to 60] | 40 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 4 | 4 | 21
  Male | 4 | 0 | 5 | 5 | 14
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 9 | 9 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alkaline Phosphatase Following 12 Weeks of Treatment
Time Frame: baseline, 12 weeks
Population: The number of participants was based on a per protocol analysis.
Measure: Median (Full Range); unit: U/L
Arm/Group | Low Dose Vancomycin | High Dose Vancomycin | Low Dose Metronidazole | High Dose Metronidazole
Number analyzed (Participants) | 7 | 8 | 7 | 6
U/L | -117 [-304 to 165] | -49 [-315 to 18] | -62 [-502 to 212] | -36 [-450 to 42]

2. Secondary Outcome: Change From Baseline in Total Bilirubin Following 12 Weeks Treatment
Time Frame: baseline, 12 weeks
Population: Per protocol analysis done
Measure: Median (Full Range); unit: mg/dl
Arm/Group | Low Dose Vancomycin | High Dose Vancomycin | Low Dose Metronidazole | High Dose Metronidazole
Number analyzed (Participants) | 7 | 8 | 7 | 6
mg/dl | -0.4 [-0.9 to 0.2] | 0.05 [-0.8 to 9.7] | -0.3 [-0.5 to 0] | 0.05 [-0.5 to 0.4]

3. Secondary Outcome: Change From Baseline in Mayo PSC Risk Score Following 12 Weeks of Treatment
Description: The Mayo PSC risk score was calculated for each patient at baseline and at 12 weeks, where Risk = 0.03 (age [years]) + 0.54 Ln (total bilirubin [mg/dL]) + 0.54 Ln (AST [IU/L]) + 1.24 (variceal bleeding) - 0.84 (albumin [g/dL]). There is no range, minimum, or maximum value but greater values indicate worse disease.
Time Frame: baseline, 12 weeks
Population: Per protocol analysis
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Low Dose Vancomycin | High Dose Vancomycin | Low Dose Metronidazole | High Dose Metronidazole
Number analyzed (Participants) | 7 | 8 | 7 | 6
units on a scale | -0.65 [-1.13 to 0.21] | -0.01 [-0.71 to 1.15] | -0.26 [-0.75 to 0.09] | -0.20 [-0.64 to 0.09]

4. Secondary Outcome: Change From Baseline in C-Reactive Protein Following 12 Weeks of Treatment
Time Frame: baseline, 12 weeks
Population: Per protocol analysis done
Measure: Median (Full Range); unit: mg/L
Arm/Group | Low Dose Vancomycin | High Dose Vancomycin | Low Dose Metronidazole | High Dose Metronidazole
Number analyzed (Participants) | 7 | 8 | 7 | 6
mg/L | -2.2 [-47.3 to 0] | 1 [-5.6 to 28.6] | -3.6 [-17.4 to 0] | 0 [-1.9 to 2.2]

ADVERSE EVENTS:
Arm/Group | Low Dose Vancomycin | High Dose Vancomycin | Low Dose Metronidazole | High Dose Metronidazole
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/8 | 3/9 | 6/9 | 8/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Vancomycin (N=8) | High Dose Vancomycin (N=9) | Low Dose Metronidazole (N=9) | High Dose Metronidazole (N=9)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (6)
anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
metallic taste (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
numbness and tingling of extremities (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
burning in eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
weight loss (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
increased fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
increased bilirubin (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
increased itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
headaches (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes